CLINICAL TRIAL: NCT02351986
Title: Effects of Cryotherapy on Inflammatory Mediators, Joint Function and Pressure Pain Threshold in Patients With Subacromial Impingement Syndrome.
Brief Title: Effects of Cryotherapy on Joint Function and Pressure Pain Threshold in Patients With Subacromial Impingement Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Aristides Leite Siqueira Junior, Master Student, Universidade Federal de Sao Carlos
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1162-2746
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Pain; Inflammation
Keywords: subacromial impingement; physical therapy; cryotherapy
MeSH Terms: conditions — Pain; Inflammation; Shoulder Impingement Syndrome | interventions — Physical Therapy Modalities

ARMS (2):
- Subacromial Impingement Syndrome (Experimental): Subjects between 18 to 45 years, with Subacromial Impingement Syndrome at least one week.
  Interventions: Procedure: physical therapy; Other: ice pack
- Control (No Intervention): Healthy subjects between 18 to 45 years.

INTERVENTIONS:
Procedure: physical therapy — A 20 minutes ice pack cryotherapy applied for 4 consecutive days
  Arms: Subacromial Impingement Syndrome
Other: ice pack
  Arms: Subacromial Impingement Syndrome

SUMMARY:
Background: Subacromial impingement syndrome (SIS) is a chronic and disabling disease, characterized by compression and mechanical abrasion of the tendons of the rotator cuff muscles, subacromial bursa and tendon of the long head of the biceps against the anterior surface of the acromion, coracoacromial ligament or the acromioclavicular joint during arm elevation movement. After the trauma, inflammatory processes initiate and may lead to loss of function when untreated. This inflammation leads the release of cytokines (IL-6, IL-10, IL-1β and TNF-α) whose acts as inflammatory mediators. Physical therapy works in treating SIS with the goal of reducing pain and inflammatory process. Cryotherapy is widely used in physical therapy by anti-inflammatory and analgesic effects, low cost, effectiveness and easy application. Objective: The aim of the study is to evaluate the effects of a cryotherapy protocol, applied on shoulder of subjects with SIS, on serum inflammatory mediators (cytokines) and local pressure pain threshold. Possible changes in function and pain will also be evaluated. Materials and Methods: 30 subjects will be selected and share in two groups, 15 healthy subjects and 15 subjects with SIS. Function assessments and quality of life will be held using the DASH and WORC questionnaires. Cryotherapy will be applied for 4 consecutive days, lasting 20 minutes without interruption through ice pack over the shoulder of SIS carriers. For the blood samples, 20ml of blood will be collected at the first and last day of the intervention, and then stored at -80 ° C.

ELIGIBILITY:
Definition: The participants will be selected from population in general and will be screened by the inclusion and exclusion criteria below:

Inclusion Criteria:

* The diagnosis for SIS will be based on a clinical examination and self-reported orthopaedic history. at least 3 positive tests of: Neer impingement test, Hawkins impingement test, Jobe test, Speed test or Gerber test, pain with passive or isometric resisted shoulder lateral rotation, pain with active shoulder elevation and pain with palpation of rotator cuff tendons.

Exclusion Criteria:

* Fracture, osteoporosis, malignancy, infection, and active inflammatory process, pregnancy, systemic illnesses, physical therapy or manual therapy treatment within 6 months prior to the evaluation, signs of complete rotator cuff tear or acute inflammation, cervicothoracic spine-related symptoms (positive cervical compression test and excessive kyphosis), scoliosis, glenohumeral instability (positive apprehension, anterior drawer, or sulcus tests), or previous upper extremity fracture or shoulder surgery.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cytokines serum levels | up to 96 hours post cryotherapy

SECONDARY OUTCOMES:
Pressure pain threshold | 72 hours pre cryotherapy and 96 hours post cryotherapy
Disabilities of the Arm, Shoulder and Hand - DASH questionnaires | 72 hours pre cryotherapy and 96 hours post cryotherapy
Western Ontario Rotator Cuff Index - WORC questionnaires | 72 hours pre cryotherapy and 96 hours post cryotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Tania Fatima Salvini, Professor, Study Director — Universidade Federal de Sao Carlos
Locations (1):
- UFSCar Physical therapy Department, São Carlos, São Paulo, Brazil